CLINICAL TRIAL: NCT03358732
Title: Effect of Intrauterine Navigation Using Intrauterine Insemination Catheter for Mock Embryo Transfer Prior to Day 3 Embryo Transfer on Pregnancy Rate: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Fahad Medical City (Other Government)
Responsible Party: Principal Investigator, Sahar Abbas Lary, Consultant, King Fahad Medical City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-460
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: The Study Focusses on Improving the Implantation Rate in IVF
Keywords: embryo transfer, mock embryo transfer, endometrial receptivity, endometrial scratching, IVF

STUDY DESIGN:
Intervention Model Description: randomized into 2 groups 1. study group had endometrial navigation using IUI catheterone day before embryo transfer control group no intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mock embryo transfer (Experimental): The patients underwent a mock embryo transfer one day before the scheduled actual transfer
  Interventions: Device: endometrial navigation one day before the embyo transfer using IUI catheter ,
- No mock embryo transfer (No Intervention): The patients did not undergo mock embryo transfer one day before the scheduled actual transfer

INTERVENTIONS:
Device: endometrial navigation one day before the embyo transfer using IUI catheter , — one day before the actual ET, the participants, in the study group, were taken into the operating room with a moderately full bladder at 10 am. The patient was placed in the lithotomy position and a sterile speculum was inserted into the vagina. The cervix was cleaned with sterile swabs and sterile water, and a mock transfer was performed using a soft catheter (Wallace Intrauterine Insemination Catheter; Sims Portex Ltd., Hythe, Kent, UK). The catheter has an outer sheet with memory , to aid insertion, and a soft inner catheter with atraumatic tip. Under ultrasound guidance, only the soft inner catheter was introduced beyond the internal cervical os till it was 0.5 cm from the fundus. It was, then, gently withdrawn out of the uterus, and the speculum was removed.
  Arms: Mock embryo transfer

SUMMARY:
Objective: To evaluate the effect of intrauterine navigation using intrauterine insemination catheter (IUI) one day prior to day 3 embryo transfer (ET) on pregnancy rate.

Design: Pilot randomized controlled study. Setting: Tertiary referral center, King Fahad Medical City. Patients: Patients who underwent ET during the period of the study after two or less in-vitro fertilization failures and fulfilled the inclusion criteria.

Interventions: Mock ETs were performed on day 2 post oocytes retrieval using intrauterine insemination catheter, followed by day 3 ET.

Main Outcome Measure: Pregnancy rate.

Key Words: embryo transfer, mock embryo transfer, endometrial receptivity, endometrial scratching, IVF.

DETAILED DESCRIPTION:
Materials and Methods Population Forty-five patients were selected for this prospective randomized control trial. It was conducted between October 2016 and October 2017 in the Reproductive Endocrinology and Infertility Medicine Department of King Fahad Medical City (KFMC).

We included nulliparous patients who were < 42 years of age with body mass index (BMI) < 30 kg/m2 and normal endometrial cavity, used fresh sperm or oocytes, had two or more embryos available for transfer on day 3 post ovum pick-up (OPU), and no more than 3 previous unsuccessful ART cycles. Patients with uterine fibroids, uterine anomalies, intra-uterine adhesions, and uterine polyps, patients with chronic diseases in the as uncontrolled diabetes or hypertension, or if the patient had difficult mock ET . patients with severe male factors for infertility requiring surgical retrieval of sperms were excluded from the study.

Ethical clearance of this study was obtained from the ethical committee of KFMC (IRB 00008644). Written informed consent was obtained from all the participants.

Stimulation Protocols Participants were assigned either to the antagonist or agonist protocol. In the agonist stimulation protocol, pituitary desensitization was achieved by using 3.75 mg leuprolide acetate (Lupron Depot, Abbott Laboratories, Chicago, USA) intramuscularly in the luteal phase of the previous cycle. The participants received 75-450 IU/d of either recombinant follicle-stimulating hormone (FSH) (Gonal-F; Serono, Munich, Germany) or highly purified human menopausal gonadotrophin (hMG) (Merional; IBSA, Lugno, Switzerland). The dosage was adjusted according to the serum E2 levels and vaginal ultrasound folliculometry. In the antagonist protocol group, 0.25 mg/d cetrorelix acetate (Cetrotide; Serono, Munich, Germany) was added on the day 5 of stimulation. When the sizes of three or more follicles became ≥16 mm, the patient was given 10,000 IU of chorionic gonadotrophin (Pregnyl; MERK, Hally, Germany) intramuscularly.

Oocyte Retrieval and Fertilization Transvaginal oocyte retrieval was scheduled 36 h after the administration of hCG and was performed under local anesthesia. Fertilization was achieved by intracytoplasmic sperm injection (ICSI). Pronuclear observation to determine fertilization was performed 16-18 h after insemination. A commercial sequential IVF medium (Cook, Eight Miles Plains, Queensland, Australia) was used for procedures involving the handling of gametes and embryos. All embryos were transferred on their respective day 3 post OPU.

Mock Embryo Transfer On day 2 post OPU, one day before the actual ET, the participants, in the study group, were taken into the operating room with a moderately full bladder at 10 am. The patient was placed in the lithotomy position and a sterile speculum was inserted into the vagina. The cervix was cleaned with sterile swabs and sterile water, and a mock transfer was performed using a soft catheter (Wallace Intrauterine Insemination Catheter; Sims Portex Ltd., Hythe, Kent, UK). The catheter has an outer sheet with memory , to aid insertion, and a soft inner catheter with atraumatic tip. Under ultrasound guidance, only the soft inner catheter was introduced beyond the internal cervical os till it was 0.5 cm from the fundus. It was, then, gently withdrawn out of the uterus, and the speculum was removed.

Embryo Transfer On the morning of ET, the patient was taken to the operating room with a moderately full bladder. To facilitate safe handling of the embryos, the operating room was connected to the embryology laboratory through a sliding door. The patient was placed in the lithotomy position and the embryos were loaded by the embryologist into the soft catheter. A maximum of two embryos were transferred per cycle. The physician then inserted the catheter into the uterus till it was approximately 1.5 cm from the fundus, and expelled the embryos. The catheter was then slowly removed from the uterus and returned to the embryologist for inspection for any remnant embryos (retained embryos for reloading), blood, or mucus.

Intravaginal progesterone (Cyclogest; 400 mg, Actavis, Devon, UK) was administered every 12 h for luteal support.

Quantitative assessment of serum ß-HCG level was performed two weeks after ET. Patients who showed high levels of serum ß-HCG were considered as pregnant and were asked to return at 6 weeks of gestation for ultrasonographic confirmation. When they returned, clinical pregnancy was determined by the observation of a gestational sac with fetal heart beat on transvaginal ultrasound. The clinical embryo implantation rate was defined as the number of gestational sacs observed at 6 weeks of gestation divided by the total number of embryos transferred.

Statistical Methods Statistical analyses were performed using SPSS (version 12.0; SPSS, Inc., Chicago, IL, USA). Results were tabulated and presented in percentages. Statistical analyses were carried out using the chi-squared test or the Fisher Exact test for categorical variables, and the unpaired two-way Student's t-test for continuous variables. A value of P ≤ 0.05 was accepted as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

We included nulliparous patients who were < 42 years of age with body mass index (BMI) < 30 kg/m2 and normal endometrial cavity, used fresh sperm or oocytes, had two or more embryos available for transfer on day 3 post ovum pick-up (OPU), and no more than 3 previous unsuccessful ART cycles

Exclusion Criteria:

Patients with uterine fibroids, uterine anomalies, intra-uterine adhesions, and uterine polyps, patients with chronic diseases in the as uncontrolled diabetes or hypertension, or if the patient had difficult mock ET . patients with severe male factors for infertility requiring surgical retrieval of sperms were excluded from the study.

-

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Biological female
Enrollment: 45 (Actual)
Dates: Start 2016-10-02 (Actual); Primary Completion 2017-10-03 (Actual); Study Completion 2017-10-03 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | 1 month
  Proportion of women with visualization of intrauterine gestation sac with positive fetal heart

CONTACTS AND LOCATIONS:
Locations (1):
- king Fahad Medical City, Riyadh, Central, Saudi Arabia